CLINICAL TRIAL: NCT07348107
Title: A Phase 1 Study of ATRA and SDK002 in Combination With Chemotherapy and Anti-PD-L1 Inhibitor in Patients With Advanced Pancreatic Ductal Adenocarcinoma.
Brief Title: ATRA and SDK002 in Combination With Chemotherapy and Anti-PD-1 Inhibitor in Patients With Advanced Pancreatic Ductal Adenocarcinoma.
Acronym: ATARI-PDAC
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Daniel Breadner (Other)
Collaborators: BeiGene (Canada) ULC (Unknown); SDK Therapeutics, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Daniel Breadner, Principal Investigator, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Organization: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ATARI-PDAC
Record Dates: First submitted 2025-12-29; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Advanced Pancreatic Ductal Adenocarcinoma
Keywords: Advanced pancreatic ductal adenocarcinoma; Metastatic; PDAC; ATRA (all-trans retinoic acid); SDK002; Tislelizumab; Gemcitabine; Nab-paclitaxel; Immune checkpoint inhibitor; Phase 1; Combination therapy; Safety and tolerability; First-line treatment; Chemotherapy; Immunotherapy
MeSH Terms: conditions — Neoplasm Metastasis | interventions — Tretinoin; Arsenic Trioxide; Gemcitabine; 130-nm albumin-bound paclitaxel; tislelizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): ATRA - 45mg/m2, oral, daily SDK002 - 10mg, oral, daily Gemcitabine - 800mg/m2, IV, Days 1, 8, 15 of a 28 day cycle Nab-paclitaxel - 125mg/m2, IV, Days 1, 8, 15 of a 28 day cycle Tislelizumab - 300mg, IV, Day 1 of a 28 day cycle
  Interventions: Drug: ATRA; Drug: Arsenic Trioxide (ATO); Drug: Gemcitabine; Drug: Nab-paclitaxel; Drug: Tislelizumab

INTERVENTIONS:
Drug: ATRA — Orally administered all-trans retinoic acid (ATRA) for up to 6 cycles in combination with chemotherapy and immunotherapy.
  Other Names: All-Trans Retinoic Acid
Drug: Arsenic Trioxide (ATO) — Orally administered SDK002 for up to 6 cycles in combination with chemotherapy and immunotherapy.
  Other Names: SDK002
Drug: Gemcitabine — Standard intravenous chemotherapy, administered per protocol.
Drug: Nab-paclitaxel — Standard intravenous chemotherapy, administered per protocol.
Drug: Tislelizumab — Anti-PD-1 immune checkpoint inhibitor, administered intravenously for up to 26 cycles.

SUMMARY:
This study is testing whether adding three drugs, All-Trans Retinoic Acid (ATRA), SDK002 (also called Arsenic Trioxide or ATO), and tislelizumab, to standard chemotherapy is safe for people with advanced pancreatic cancer. Advanced pancreatic cancer means the cancer has spread or cannot be removed with surgery. The study will also look at whether this treatment combination may help people live longer.

Participants will receive standard chemotherapy drugs, gemcitabine and nab-paclitaxel, together with ATRA, SDK002, and tislelizumab. ATRA is related to vitamin A and may affect how cancer cells grow. SDK002 is a drug used to treat sine cancers and may help other treatments work better. Tislelizumab is an immunotherapy drug, which helps the immune system recognize and attack cancer cells. This is a phase 1 study, which means the main goal is to test safety and side effects. All participants receive the same treatment, and both the study doctors and participants know which drugs are being given.

DETAILED DESCRIPTION:
This is a Phase 1, open-label, single center study to evaluate the safety of ATRA and SDK002 when given with gemcitabine, nab-paclitaxel and tislelizumab in participants with previously untreated, unresectable/metastatic pancreatic ductal adenocarcinoma. The enrolment target is 6 to 10 participants over 6 months.

An initial safety run-in will cap the gemcitabine dose at 800 mg/m2 in addition to standard dose ATRA, SDK002, nab-paclitaxel and tislelizumab. If the first 3 participants receiving 800 mg/m2 gemcitabine at each C1 administration do not experience grade 3+ AEs related to gemcitabine, the Steering Committee (SC) will review the data and may approve the option to escalate gemcitabine to the standard maximum dose of 1000 mg/m2 at C2D1 for subsequent participants. Safety data for participants treated at 1000 mg/m2 will be reviewed at each applicable SC meeting. Once a safe dose has been established, accrual will halt and the SC will establish the maximum dose of gemcitabine permitted in a future Phase 2 study.

After a screening period of up to 28 days, each participant will receive orally administered ATRA and SDK002 for a maximum of 6 cycles in combination with gemcitabine and nab-paclitaxel (until progression or unacceptable toxicity), and tislelizumab (for a maximum of 2 years or until progression or unacceptable toxicity). After treatment, each participant will be followed for 2 years, or until recurrence/death is documented, whichever comes first.

Participants may continue both ATRA and SDK002 while on at least one chemotherapy agent (gemcitabine or nab-paclitaxel) and/or immune checkpoint inhibitor (tislelizumab). Participants who permanently discontinue both the immune checkpoint inhibitor and the entire chemotherapy regimen must stop ATRA and SDK002, at which point the participant will be considered off protocol treatment.

All participants are highly recommended to have fresh tumor biopsies collected between C2 and C3. If a participant withdraws consent for this biopsy they will not be removed from the study, but should only be accrued if their initial intent is to undergo an on treatment biopsy.

Participants will return for a Safety Follow-up Visit 28 (± 7) days after the end of the last cycle. Participants who experience disease progression/relapse will enter Survival Follow-up and be contacted every 3 months after the end of the last cycle date for late onset immune related AEs, then every 6 months until death.

Safety will be assessed by AEs, clinical laboratory evaluation (serum chemistry, hematology, coagulation, and urinalysis), physical examination, vital signs measurements, ECGs (including QTc interval), and ECOG performance status.

Exploratory endpoints will include assessments of correlative tissue and blood-based biomarkers associated with drug target engagement, drug synergy and treatment response or resistance.

ELIGIBILITY:
Inclusion Criteria

* Participants must have previously untreated unresectable/ metastatic PDAC, without plans for a curative surgery, previous neoadjuvant therapy with 5-FU based therapy is permitted but neoadjuvant gemcitabine-based therapy must have been completed at least 6-months prior to enrollment without documented progression while on gemcitabine. Unresectable PDAC is determined based surgical assessment deeming that curative resection is not foreseeable or appropriate.
* Participants should have adequate archival tissue (from primary or metastatic tumour) available and must have provided informed consent for the release of this tissue. For potential participants who do not have adequate residual tissue or a biopsy which was only suspicious for adenocarcinoma approval from the sponsor prior to enrollment is required.
* Participants must be ≥ 18 years of age.
* Participants must have an ECOG performance status of 0 to 2.
* Participants must have a life expectancy of 3 months or longer.
* Laboratory requirements (must be done within 7 days prior to enrollment):
* Absolute neutrophils: ≥ 1.5 × 109/L (without granulocyte colony-stimulating factor support within 2 weeks prior to the first study treatment)
* Hemoglobin: ≥ 90 × 109/L
* Platelets: ≥ 100 × 109/L
* Bilirubin: < 1.5 × ULN (Note: Exceptions may be made if confirmed diagnosis of Gilberts (< 3 × ULN); ≤ 5.0 × ULN if participant has liver metastases or partial biliary obstruction post stenting or drainage and felt to be stable
* AST and ALT: < 2.5 × ULN; ≤ 5.0 × ULN if participant has liver metastases or partial biliary obstruction post stenting or drainage and felt to be stable
* ALP: < 2.5 × ULN; ≤ 5.0 × ULN if participant has liver metastases or partial biliary obstruction post stenting or drainage and felt to be stable
* Serum creatinine and creatinine clearance: ≥ 45 mL/min; (Note: Creatinine clearance to be measured directly by 24-hour urine sampling or as calculated by Cockcroft and Gault equation below:

Females: GFR = 1.04 × [140-age] × weight in kg / serum creatinine in μmol/L

Males: GFR = 1.23 × [140-age] × weight in kg / serum creatinine in μmol/)

* Participants must be able to swallow oral medications and have no known gastrointestinal disorders that may interfere with absorption (such as malabsorption).
* Patients must have received no prior systemic therapy in the first-line setting for unresectable/metastatic disease.
* Prior chemotherapy: prior chemotherapy in the adjuvant/neoadjuvant setting is allowed provided > 6 months from last chemotherapy at time of enrolment for gemcitabine-based therapies, no time restrictions for 5-FU based therapies; patients must have had recovered (to grade 1 or better) from all reversible toxicity related to prior chemotherapy or systemic therapy.
* Radiation: Prior external beam radiation is permitted provided a minimum of 28 days (4 weeks) have elapsed between the last dose of radiation and date of enrollment. Exceptions include low-dose, non-myelosuppressive radiotherapy to sites outside of the primary disease such as palliative radiation to bone metastases. Concurrent radiotherapy is not permitted.
* Surgery: Previous surgery is permitted provided that a minimum of 21 days (3 weeks) have elapsed between any major surgery and date of enrollment, and that wound healing has occurred. Stenting, percutaneous cholecystostomy, and endoscopies are permitted.
* Interventional Radiology: Prior radioembolization is permitted up to 4 weeks prior to enrolment. Interventional pain control such as celiac axis block allowed prior to treatment.
* Participant consent must be appropriately obtained in accordance with applicable local and regulatory requirements. Each participant must sign a consent form prior to screening (if applicable)/enrollment in the trial to document their willingness to participate.
* Participants must be accessible for treatment and follow up. Participants enrolled in this trial must be treated and followed at the participating center. Investigators must assure themselves the participants enrolled in this trial will be available for complete documentation of the treatment, AEs, and follow-up.
* Participants of childbearing potential (WOCBP) must agree to use a highly effective contraceptive method. A woman is considered to be of "childbearing potential" if she has had menses at any time in the preceding 12 consecutive months.
* WOCBP will have a pregnancy test to determine eligibility as part of the pre-study evaluation; this may include an ultrasound to rule-out pregnancy if a false-positive is suspected. For example, when beta-human chorionic gonadotropin (hCG) is elevated from a possible tumour source. Participants will be considered eligible if an ultrasound is negative for pregnancy.

Male participants should also refrain from donating sperm during the study and for 6 months after the last dose of study treatment.

-Women must refrain from breastfeeding while on treatment.

Exclusion Criteria

* Participants with any medical condition that would impair the administration of oral agents including significant bowel resection, inflammatory bowel disease or uncontrolled vomiting.
* Participants with a history of other malignancies, except adequately treated non-melanoma skin cancer and low-grade prostate cancer, curatively treated in-situ cancer of the cervix, or other solid tumours curatively treated with no evidence of disease for > 2 years.
* Participants may not receive concurrent treatment with other anti-cancer therapy (other than bone-targeted therapy, GnRH agonist/antagonist, or adjuvant tamoxifen and aromatase inhibitors if already taking and stable) or investigational agents while on protocol therapy. Concurrent use of hormonal therapy for non-cancer-related conditions (e.g., hormone replacement therapy) is acceptable.
* Participants with history of allogeneic organ transplantation.
* Participants with active autoimmune or inflammatory disorders (including inflammatory bowel disease [e.g., colitis or Crohn's disease], systemic lupus erythematosus, Sarcoidosis syndrome, or granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc.]) that has required systemic treatment in past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
* The following autoimmune are exceptions to this criterion: 1) participants with vitiligo or alopecia; 2) participants with hypothyroidism (e.g., following Hashimoto syndrome) stable on hormone replacement; 3) participants with any chronic skin condition that does not require systemic therapy; 4) participants with celiac disease controlled by diet alone; 5) participants without an active disease in the last 5 years may be included but only after consultation with the principal investigator.
* Current or prior use of immunosuppressive medications within 14 days before first drug dose.
* The following are exceptions to this criterion: 1) intranasal, inhaled, or topical steroids or local steroid injections (e.g., intra-articular injection); 2) systemic corticosteroids at physiologic doses not to exceed 10 mg/day of prednisone or its equivalent; 3) steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication) or steroids a single oral dose are permitted
* History of active primary immunodeficiency.
* Participants who have received growth factors within 28 days prior to initiation of dosing of ATRA and SDK002.
* Primary prophylaxis not allowed, but secondary prophylaxis is permitted.
* Participant has known active, uncontrolled HIV, or hepatitis B or C infection.
* Participants with undetectable viral load are eligible.
* Participants with serious illnesses which would not permit the participant to be managed according to the protocol.
* Uncontrolled intercurrent illness includes but is not limited to: clinically active diverticulitis, intra-abdominal abscess, GI obstruction, abdominal carcinomatosis, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, uncontrolled cardiac arrhythmia, active interstitial lung disease (ILD), serious chronic gastrointestinal conditions associated with diarrhea, or psychiatric illness/social situations that would limit compliance with study requirement, substantially increase the risk of incurring AEs, or compromise the ability of the participant to give written informed consent.
* Participant deemed by the investigator to be at high cardiovascular risk, specifically including, but not limited to, recent coronary stenting or myocardial infarction in the 6 months before screening, or QTc ≥ 490 ms for males or ≥ 470 ms for females.
* Participants with pre-existing sensory neuropathy > grade 1.
* Participants with history of central nervous system metastases or spinal cord compression unless they have received treatment, are clinically stable and do not require corticosteroids.
* Participants with symptomatic ascites or pleural effusion. Participants who are clinically stable following treatment for these conditions (including therapeutic thoracentesis or paracentesis) are eligible.
* Participants are not eligible if they have a known hypersensitivity to the study drug(s) or their components.
* Major surgical procedure within 28 days before the first dose of study treatment.
* Participants who have received prior immune-mediated therapy, including, but not limited to, other anti-PD-1, anti PD-L1, or anti CTLA-4.
* Participant is taking any additional cytotoxic anti-cancer medications, other prohibited concurrent medication, including vitamin A supplements, isotretinoin, and is unwilling to stop use prior to and during the trial.
* Participant has received a live vaccine within 4 weeks before receiving their first dose of study treatment.
* Participant is unwilling or unable to comply with study procedures, as assessed by the Principal Investigator.
* Is pregnant, breastfeeding, or is of reproductive potential and unwilling to comply with contraceptive requirements as described in Appendix 5.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2026-02-15 (Estimated); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events as Assessed by CTCAE v5.0 | Up to 6 months.
  Safety will be evaluated by the incidence of adverse events (AEs), including serious adverse events (SAEs), grade 3 and 4 adverse events, adverse events of all grades, and adverse events leading to the discontinuation of study medication. Adverse events will be graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE), version 5.0. Safety outcomes will be analyzed using descriptive analyses, including the number and percentage of participants with AEs, SAEs, deaths, adverse events leading to treatment discontinuation, and adverse events by severity and relatedness. Adverse events will be summarized by system organ class and preferred term using the Medical Dictionary for Regulatory Activities (MedDRA). Clinically significant changes in vital signs and clinical laboratory results will be summarized descriptively, and shift tables will be provided showing change in CTCAE grade from baseline to worst post-baseline grade.

SECONDARY OUTCOMES:
6-Month Progression-Free Survival Rate | 6 months.
  The 6-month progression-free survival (PFS) rate is defined as the proportion of participants who remain alive and progression-free at 6 months from the start of study treatment. Tumour progression will be assessed by the site radiologist and/or investigator using iRECIST v1.1 criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Breadner, Principal Investigator — London Health Sciences Centre Research Institute
Locations (1):
- Verspeeten Family Cancer Centre, London, Ontario, Canada